CLINICAL TRIAL: NCT03618056
Title: A Phase 1b Open Label Clinical Trial to Evaluate HIV-1 Neutralization Antibody Breadth in Response to HIV gp120 Protein Vaccine in HIV-uninfected Adults With Quiescent Systemic Lupus Erythematosus
Brief Title: Evaluating HIV-1 Neutralization Antibody Breadth in Response to HIV gp120 Protein Vaccine in HIV-uninfected Adults With Quiescent Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: HVTN 121; 38162 (Registry Identifier: DAIDS-ES Registry Number)
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Results first posted 2021-12-29 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: HIV Infections; Systemic Lupus Erythematosus
MeSH Terms: conditions — HIV Infections; Lupus Erythematosus, Systemic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AIDSVAX® B/E (Experimental): Participants will receive 600 mcg/mL of AIDSVAX® B/E at Months 0, 1, and 6.
  Interventions: Biological: AIDSVAX® B/E

INTERVENTIONS:
Biological: AIDSVAX® B/E — Administered by intramuscular injection

SUMMARY:
The purpose of this study is to evaluate the breadth and potency of HIV-1 neutralizing antibody (nAb) responses and examine the safety and tolerability of an HIV gp120 protein vaccine (AIDSVAX® B/E) in HIV-uninfected adults diagnosed with Systemic Lupus Erythematosus (SLE) who have stable disease.

DETAILED DESCRIPTION:
This study will evaluate the breadth and potency of HIV-1 neutralizing antibody (nAb) responses and examine the safety and tolerability of an HIV gp120 protein vaccine (AIDSVAX® B/E) in HIV-uninfected adults diagnosed with Systemic Lupus Erythematosus (SLE) who have stable disease.

All participants will receive 600 mcg/mL of AIDSVAX® B/E at Months 0, 1, and 6.

Study visits will occur at Months 0, 0.25, 0.5, 1, 1.25, 1.5, 3, 6, 6.25, 6.5, 7.5, 8.5, and 12. Visits may include physical examinations, blood and urine collection, pregnancy testing, HIV testing, risk reduction counseling, assessments, and questionnaires.

ELIGIBILITY:
Inclusion Criteria:

General and Demographic Criteria

* Age of 18 to 50 years
* Weight greater than 110 pounds
* Meets American College of Rheumatology (ACR) criteria for the classification of SLE with serologic evidence of disease including a positive test for antinuclear antibodies at a titer of 1:640 or greater, or the presence of a positive test for antibodies to double-strand DNA (dsDNA), or the presence of anti-Sm, anti-RNP, or anti-Ro antibodies, as documented by medical records and as assessed by a rheumatologist or designee.
* Currently taking hydroxychloroquine for SLE and for at least 6 months prior to enrollment
* Access to a participating HIV Vaccine Trials Network (HVTN) clinical research site (CRS) and willingness to be followed for the planned duration of the study
* Ability and willingness to provide informed consent
* Allows ongoing access to medical records pertaining to their rheumatologic disease
* Assessment of understanding: volunteer demonstrates understanding of this study; completes a questionnaire prior to first vaccination with verbal demonstration of understanding of all questionnaire items answered incorrectly
* Agrees not to enroll in another study of an investigational research agent before the last required protocol clinic visit

HIV-Related Criteria:

* Willingness to receive HIV test results
* Willingness to discuss HIV infection risks and amenable to HIV risk reduction counseling.
* Assessed by the clinic staff as being at "low risk" for HIV infection and committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit (see protocol for more information)

Laboratory Inclusion Values

Hemogram/Complete blood count (CBC)

* Hemoglobin greater than or equal to 11.0 g/dL for volunteers who were assigned female sex at birth, greater than or equal to 12.0 g/dL for volunteers who were assigned male sex at birth.
* White blood cell count equal to 2,500 to 12,000 cells/mm^3
* Total lymphocyte count greater than or equal to 800 cells/mm^3
* Remaining differential either within institutional normal range or with site physician approval
* Platelets equal to 100,000 to 550,000/mm^3

Chemistry

* Chemistry panel: alanine amino transferase (ALT) and aspartate aminotransferase (AST) less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to institutional upper limit of normal.

Virology

* Negative HIV-1 and -2 blood test: volunteers must have a negative US Food and Drug Administration (FDA)-approved enzyme immunoassay (EIA) within 56 days prior to enrollment.
* Negative Hepatitis B surface antigen (HBsAg) within 56 days prior to enrollment
* Negative anti-Hepatitis C virus antibodies (anti-HCV), or negative HCV polymerase chain reaction (PCR) if the anti-HCV is positive within 56 days prior to enrollment

Urine

* Normal urine by urinalysis:

  * Negative urine glucose, and
  * Negative or trace urine protein, and
  * Red blood cell (RBC) levels within institutional normal range, and
  * No RBC casts

Reproductive Status

* Volunteers who were assigned female sex at birth: negative serum or urine beta human chorionic gonadotropin (β-HCG) pregnancy test in accordance with local regulatory requirements, performed prior to vaccination on the day of initial vaccination. Persons who are NOT of reproductive potential due to having undergone total hysterectomy or bilateral oophorectomy (verified by medical records), are not required to undergo pregnancy testing.
* Reproductive status: A volunteer who was assigned female sex at birth must:

  * Agree to use effective contraception for sexual activity that could lead to pregnancy from at least 21 days prior to enrollment through the last required protocol clinic visit. Effective contraception is defined as using the following methods:

    * Condoms (male or female) with or without a spermicide,
    * Diaphragm or cervical cap with spermicide,
    * Intrauterine device (IUD),
    * Hormonal contraception, or
    * Any other contraceptive method approved by the HVTN 121 Protocol Safety Review Team (PSRT)
    * Successful vasectomy in any partner assigned male sex at birth (considered successful if a volunteer reports that a male partner has [1] documentation of azoospermia by microscopy, or [2] a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity postvasectomy);
  * Or not be of reproductive potential, such as having reached menopause (no menses for 1 year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation;
  * Or be sexually abstinent.
* Volunteers who were assigned female sex at birth must also agree not to seek pregnancy through alternative methods, such as artificial insemination or in vitro fertilization until after the last required protocol clinic visit

Exclusion Criteria:

General

* Blood products received within 120 days before first vaccination
* Investigational research agents not used to treat SLE received within 30 days before first vaccination (additional exclusions may apply, see criteria below)
* Intent to participate in another study of an investigational research agent or any other study that requires non-HVTN HIV antibody testing during the planned duration of the HVTN 121 study
* Pregnant or breastfeeding
* Active duty and reserve US military personnel

SLE status. The following criteria must be verified by a rheumatologist or designee

* Currently with active lupus as defined by a Systemic Lupus Erythematosus Disease Activity Index (SELENA-SLEDAI) greater than 4 (see protocol for more information).
* Documented SLEDAI score of greater than 20 in medical record at any time indicating severe activity, or evidence of moderate disease activity (SELENA-SLEDAI greater than 6) within the last six months, (see protocol for more information).
* Has had a condition listed on the Systemic Lupus International Collaborating Clinics/American College of Rheumatology Damage Index (SLICC/ACR DI) or has had an increase in the SLICC/ACR D1 score within the last 12 months other than cataracts, premature ovarian failure or diabetes mellitus with approval of the PSRT http://www.clinexprheumatol.org/article.asp?a=2697
* A history of central nervous system (CNS) disease
* Thrombotic event within the past 12 months in association with confirmed antiphospholipid antibody
* A history of renal disease (SLE-related renal injury) confirmed by prior biopsy, active urine sediment, or proteinuria
* Prednisone dose greater than 10 mg/day for more than 6 months within the past year
* Administration of anti-B-cell therapy (rituximab or belimumab) or any investigational research agents used to treat SLE within the preceding 2 years
* Administration of cyclophosphamide within the preceding year; or administration of mycophenolate mofetil within the last 6 months; or administration of methotrexate, leflunomide, or azathioprine within the last 3 months
* Administration of any investigational immunosuppressant medication within the last year
* Administration of other immunosuppressive medications not listed above, with the exception of topical steroids, topical immunosuppressives (eg, cyclosporine, FK506), or ophthalmic immunosuppressives (eg, steroids, cyclosporine), within 6 months before first vaccination, unless approved by the HVTN 121 PSRT

Vaccines and other Injections

* HIV vaccine(s) received in a prior HIV vaccine trial. For volunteers who have received control/placebo in an HIV vaccine trial, the HVTN 121 PSRT will determine eligibility on a case-by-case basis.
* Non-HIV experimental vaccine(s) received within the last 5 years in a prior vaccine trial. Exceptions may be made by the HVTN 121 PSRT for vaccines that have subsequently undergone licensure by the FDA. For volunteers who have received control/placebo in an experimental vaccine trial, the HVTN 121 PSRT will determine eligibility on a case-by-case basis. For volunteers who have received an experimental vaccine(s) greater than 5 years ago, eligibility for enrollment will be determined by the HVTN 121 PSRT on a case-by-case basis.
* Vaccines received within 30 days before first study vaccination or scheduled within 30 days after injection (eg, influenza, tetanus, pneumococcal, Hepatitis A or B, measles, mumps, and rubella [MMR]; oral polio vaccine [OPV]; varicella; yellow fever)
* Allergy treatment with antigen injections within 30 days before first vaccination or that are scheduled within 14 days after first vaccination

Immune System

* Serious adverse reactions to vaccines or to vaccine components (such as yeast protein, amorphous aluminum hydroxyphosphate sulfate, L-histidine, polysorbate 80, sodium borate), including history of anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. (Not excluded from participation: a volunteer who had a nonanaphylactic adverse reaction to pertussis vaccine as a child.)
* Immunoglobulin received within 60 days before first vaccination
* Immunodeficiency, such as common variable immunodeficiency

Clinically significant medical conditions

* Ongoing bleeding or hemorrhage (excluding menstruation), or any subject on anticoagulant therapy
* Clinically significant medical condition, physical examination findings, clinically significant abnormal laboratory results, or past medical history with clinically significant implications for current health, other than SLE and its manifestations. A clinically significant condition or process includes but is not limited to:

  * A process that would affect the immune response,
  * A process that would require medication that affects the immune response,
  * Any contraindication to repeated injections or blood draws,
  * A condition that requires active medical intervention or monitoring to avert grave danger to the volunteer's health or well-being during the study period,
  * A condition or process for which signs or symptoms could be confused with reactions to vaccine, or
  * Any condition specifically listed among the exclusion criteria below.
* Any medical, psychiatric, occupational, or other condition that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a volunteer's ability to give informed consent
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with psychoses within the past 3 years, ongoing risk for suicide, or history of suicide attempt or gesture within the past 3 years.
* Current anti-tuberculosis (TB) prophylaxis or therapy
* Asthma exclusion criteria: Asthma other than mild, well-controlled asthma. (Symptoms of asthma severity as defined in the most recent National Asthma Education and Prevention Program (NAEPP) Expert Panel report). Exclude a volunteer who:

  * Uses a short-acting rescue inhaler (typically a beta 2 agonist) daily, or
  * Uses moderate/high dose inhaled corticosteroids, or
  * In the past year has either of the following:

    * Greater than 1 exacerbation of symptoms treated with oral/parenteral corticosteroids;
    * Needed emergency care, urgent care, hospitalization, or intubation for asthma.
* Uncontrolled diabetes mellitus, Hb A1C greater than 7.0. (not excluded: history of isolated gestational diabetes.)
* Uncontrolled hypertension:

  * If a person has a history of hypertension, or is found to have elevated blood pressure or hypertension during screening, exclude for blood pressure that is not well controlled. Well-controlled blood pressure is defined as consistently less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic, with only isolated, brief instances of higher readings, which must be less than or equal to 150 mm Hg systolic and less than or equal to 100 mm Hg diastolic. For these volunteers, blood pressure must be less than or equal to 140 mm Hg systolic and less than or equal to 90 mm Hg diastolic at enrollment.
  * If a person has NOT been found to have elevated blood pressure or hypertension during screening or previously, exclude for systolic blood pressure greater than or equal to 150 mm Hg at enrollment or diastolic blood pressure greater than or equal to 100 mm Hg at enrollment.
* Bleeding disorder diagnosed by a doctor (eg, factor deficiency, coagulopathy, or platelet disorder requiring special precautions)
* Malignancy (not excluded from participation: Volunteer who has had malignancy excised surgically and who, in the investigator's estimation, has a reasonable assurance of sustained cure, or who is unlikely to experience recurrence of malignancy during the period of the study)
* Seizure disorder: History of seizure(s) within past three years. Also exclude if volunteer has used medications in order to prevent or treat seizure(s) at any time within the past 3 years.
* Asplenia: any condition resulting in the absence of a functional spleen (not excluded: splenectomy for splenic trauma)
* History of hereditary angioedema, acquired angioedema, or idiopathic angioedema.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2020-07-17 (Actual); Study Completion 2020-07-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: M. Anthony Moody, Study Chair — Duke University; Paul Goepfert, Study Chair — University of Alabama at Birmingham
Locations (1):
- Duke Human Vaccine Institute CRS, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AIDSVAX® B/E
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Response Rates of nAb Responses to the Vaccine Strains and a Global Panel of Heterologous Env-pseudotyped Viruses
Description: Assessed by TZM-bl assay
Time Frame: Measured through Month 6.5
Population: Data have not been collected for this Outcome and cannot be reported. This is due to the enrollment of only one participant in this study and the subsequent lack of ability to draw conclusions that would answer the study objectives from data from one participant.
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 0

2. Primary Outcome: Change in Magnitude of nAb Responses to the Vaccine Strains and a Global Panel of Heterologous Env-pseudotyped Viruses
Description: Assessed by TZM-bl assay
Time Frame: Measured through Month 6.5
Population: as for outcome 1
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 0

3. Primary Outcome: Breadth of nAb Responses to the Vaccine Strains and a Global Panel of Heterologous Env-pseudotyped Viruses
Description: Assessed by TZM-bl assay
Time Frame: Measured through Month 6.5
Population: as for outcome 1
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 0

4. Primary Outcome: Number of Participants With Local Reactogenicity Signs and Symptoms, Stratified by Severity
Description: Graded according to the Division of AIDS (DAIDS) Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July, 2017. The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured for seven days through participant's last vaccination at Month 0,1,and 6
Measure: Count of Participants; unit: Participants
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 1
Participants
  Erythema: None | 0
  Erythema: Mild | 1
  Erythema: Moderate | 0
  Erythema: Severe | 0
  Erythema: Life-threatening | 0
  Induration: None | 0
  Induration: Mild | 1
  Induration: Moderate | 0
  Induration: Severe | 0
  Induration: Life-threatening | 0
  Pain/Tenderness: None | 0
  Pain/Tenderness: Mild | 1
  Pain/Tenderness: Moderate | 0
  Pain/Tenderness: Severe | 0
  Pain/Tenderness: Life-threatening | 0

5. Primary Outcome: Number of Participants With Systemic Reactogenicity Signs and Symptoms, Stratified by Severity
Description: Graded according to the DAIDS Table for Grading the Severity of Adult and Pediatric Adverse Events, Corrected Version 2.1, July, 2017. The maximum grade observed for each symptom over the time frame is presented.
Time Frame: Measured for seven days through participant's last vaccination at Month 0,1,and 6
Measure: Count of Participants; unit: Participants
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 1
Participants
  Fever: None | 1
  Fever: Mild | 0
  Fever: Moderate | 0
  Fever: Severe | 0
  Fever: Life-threatening | 0
  Malaise/Fatigue: None | 1
  Malaise/Fatigue: Mild | 0
  Malaise/Fatigue: Moderate | 0
  Malaise/Fatigue: Severe | 0
  Malaise/Fatigue: Life-threatening | 0
  Myalgia: None | 1
  Myalgia: Mild | 0
  Myalgia: Moderate | 0
  Myalgia: Severe | 0
  Myalgia: Life-threatening | 0
  Headache: None | 0
  Headache: Mild | 1
  Headache: Moderate | 0
  Headache: Severe | 0
  Headache: Life-threatening | 0
  Nausea: None | 1
  Nausea: Mild | 0
  Nausea: Moderate | 0
  Nausea: Severe | 0
  Nausea: Life-threatening | 0
  Chills: None | 1
  Chills: Mild | 0
  Chills: Moderate | 0
  Chills: Severe | 0
  Chills: Life-threatening | 0
  Arthralgia: None | 1
  Arthralgia: Mild | 0
  Arthralgia: Moderate | 0
  Arthralgia: Severe | 0
  Arthralgia: Life-threatening | 0

6. Primary Outcome: Number of Participants With Adverse Events, by Relationship to the Study Product
Description: AEs categorized by Medical Dictionary for Regulatory Activities (MedDRA) System Organ Class, and MedDRA Preferred Term. For participants reporting multiple AEs over the time frame, the maximum relationship is counted.
Time Frame: Measured through Month 12
Measure: Count of Participants; unit: Participants
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 1
Participants
  Related | 0
  Not Related | 1
  No AEs reported | 0

7. Primary Outcome: Number of Participants With SLE Disease Activity and Functional Status Scores, by Score and Study Day
Description: As assessed by Safety of Estrogens in Lupus Erythematosus National Assessment-SLE Disease Activity Index (SELENA-SLEDAI) and Routine Assessment of Patient Index Data (RAPID3). The SELENA-SLEDAI is used to assess disease activity across nine organ systems within 10 days prior up to and including the day of study visit. The SELENA-SLEDAI is reported as a a weighted composite score with a range from 0 (no evidence of disease; best outcome) to 105 (extremely severe disease). The RAPID3 is a pooled index of the 3 patient-reported American College of Rheumatology rheumatoid arthritis (RA) Core Data Set measures: function, pain, and patient global estimate of status. Each of the 3 individual measures is scored 0 to 10, for a total of 30. Disease severity was classified on the basis of RAPID3 scores: >12 = high severity; 6.1-12 = moderate; 3.1-6 = low; < or =3 = near remission (best outcome).
Time Frame: Measured at all study visits completed in person through Month 12. Per protocol, the assessments were administered at Screening, Day 0 (date of first vaccination), Day 7, Day 14, Day 35, Day 42, Day 84, Day 168, Day 175, Day 182, Day 238, and Day 364.
Measure: Count of Participants; unit: Participants
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 1
Participants
  SELENA-SLEDAI score 0 at screening | 1
  SELENA-SLEDAI score 0 at Day 0 | 1
  SELENA-SLEDAI score 0 at Day 7 | 1
  SELENA-SLEDAI score 0 at Day 14 | 1
  SELENA-SLEDAI score 0 at Day 28 | 1
  SELENA-SLEDAI score 0 at Day 35 | 1
  SELENA-SLEDAI score 0 at Day 42 | 1
  SELENA-SLEDAI score 0 at Day 84 | 1
  SELENA-SLEDAI score 0 at Day 168 | 1
  SELENA-SLEDAI score 0 at Day 175 | 1
  SELENA-SLEDAI score 0 at Day 182 | 1
  SELENA-SLEDAI score not done at Day 238 | 1
  SELENA-SLEDAI score 0 at Day 364 | 1
  Rapid 3 Score of Near Remission (NR) at screening | 1
  Rapid 3 Score of Near Remission (NR) at Day 1 | 1
  Rapid 3 Score of Near Remission (NR) at Day 7 | 1
  Rapid 3 Score of Near Remission (NR) at Day 14 | 1
  Rapid 3 Score of Near Remission (NR) at Day 21 | 1
  Rapid 3 Score of Near Remission (NR) at Day 35 | 1
  Rapid 3 Score of Near Remission (NR) at Day 42 | 1
  Rapid 3 Score of Near Remission (NR) at Day 84 | 1
  Rapid 3 Score of Near Remission (NR) at Day 168 | 1
  Rapid 3 Score of Near Remission (NR) at Day 175 | 1
  Rapid 3 Score of Near Remission (NR) at Day 182 | 1
  Rapid 3 Score not assessed at Day 238 | 1
  Rapid 3 Score of Near Remission (NR) at Day 365 | 1

8. Secondary Outcome: Changes in Somatic Hypermutation in Participants With SLE Compared With Historical Controls
Description: Measured by flow cytometry
Time Frame: Measured through Month 6.5
Population: as for outcome 1
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 0

9. Secondary Outcome: Change in Length of Antibody Binding Loops and Germline Gene Usage in Participants With SLE Compared With Historical Controls
Description: Measured by flow cytometry
Time Frame: Measured through Month 6.5
Population: as for outcome 1
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in NAb Responses to Viruses With Altered Glycosylation, Indicative of bnAb Precursors
Description: Assessed by TZM-bl assay
Time Frame: Measured through Month 6.5
Population: as for outcome 1
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Vaccine-induced Immune Activation
Description: Assessed by serum cytokine analysis and B and T cell phenotyping, as well as expression of Treg and Tfh markers
Time Frame: Measured through Month 6.25
Population: as for outcome 1
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 0

12. Secondary Outcome: Change in Response Rate of HIV-1-Specific IgG Binding Antibodies
Description: Assessed by Binding Antibody Multiplex Assay (BAMA)
Time Frame: Measured through Month 6.5
Population: as for outcome 1
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 0

13. Secondary Outcome: Change in Magnitude of HIV-1-Specific IgG Binding Antibodies
Description: Assessed by BAMA
Time Frame: Measured through Month 6.5
Population: as for outcome 1
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 0

14. Secondary Outcome: Change in Specificity of Antibody Responses
Description: Assessed by epitope mapping of functional and binding antibodies
Time Frame: Measured through Month 6.5
Population: as for outcome 1
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 0

15. Secondary Outcome: Change in Response Rate of Env-specific CD4+ T Cells
Description: Measured by intracellular cytokine staining (ICS)
Time Frame: Measured through Month 6.5
Population: as for outcome 1
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 0

16. Secondary Outcome: Change in Magnitude of Env-specific CD4+ T Cells
Description: Measured by ICS
Time Frame: Measured through Month 6.5
Population: as for outcome 1
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 0

17. Secondary Outcome: Change in Polyfunctionality of Env-specific CD4+ T Cells
Description: Measured by ICS
Time Frame: Measured through Month 6.5
Population: as for outcome 1
Arm/Group | AIDSVAX® B/E
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Data were collected for 12 months of study participation.
Arm/Group | AIDSVAX® B/E
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AIDSVAX® B/E (N=1)
Urinary tract infection (Infections and infestations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03618056/Prot_SAP_001.pdf
  • Informed Consent Form (2018-09-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT03618056/ICF_000.pdf